CLINICAL TRIAL: NCT01530763
Title: A Multicenter, Randomized, Observer-Blinded, Active-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Ceftaroline Versus Ceftriaxone in Pediatric Subjects With Community-acquired Bacterial Pneumonia Requiring Hospitalization
Brief Title: Safety and Efficacy Study of Ceftaroline Versus a Comparator in Pediatric Subjects With Community Acquired Bacterial Pneumonia (CABP)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P903-31
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Infections; Community Acquired Pneumonia
Keywords: Infections; Pediatrics; Teflaro; cephalosporin
MeSH Terms: conditions — Infections; Community-Acquired Pneumonia | interventions — Ceftaroline; Ceftriaxone; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftaroline fosamil (Experimental)
  Interventions: Drug: Ceftaroline fosamil; Drug: amoxicillin clavulanate
- Ceftriaxone (Active Comparator)
  Interventions: Drug: Ceftriaxone; Drug: amoxicillin clavulanate

INTERVENTIONS:
Drug: Ceftaroline fosamil — Treatment Group 1:
  Drug: Ceftaroline fosamil Children ≥ 6 months: IV ceftaroline fosamil 12 mg/kg for subjects weighing ≤ 33 kg or 400 mg for subjects weighing > 33 kg will be infused over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour)
  Children < 6 months: Ceftaroline fosamil 8 mg/kg over 60 (± 10) minutes q8h (± 1 hour)
  Other Names: Teflaro; PPI-0903; TAK-599; TAK599; PPI0903
  Arms: Ceftaroline fosamil
Drug: Ceftriaxone — Treatment group 2:
  75 mg/kg/day up to 4 g/day IV in equally divided doses, each infused over 30 (± 10) minutes q12hr (± 2 hours)
  Arms: Ceftriaxone
Drug: amoxicillin clavulanate — Oral Switch for Treatment Groups 1 and 2:
  PO amoxicillin clavulanate 90 mg/kg/day divided q12h in subjects with infections due to susceptible organisms on or after Study Day 4 (a minimum of 7 IV doses required if randomized to ceftaroline.)

SUMMARY:
This is a study of safety and effectiveness of ceftaroline fosamil in children with Community Acquired Bacterial Pneumonia receiving antibiotic therapy in the hospital.

DETAILED DESCRIPTION:
To evaluate safety, effectiveness, pharmacokinetics and tolerance of ceftaroline fosamil in children who are initially hospitalized with Community Acquired Bacterial Pneumonia (CABP)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 2 months to < 18 years old.
* Presence of CABP requiring hospitalization and IV antibacterial therapy

Exclusion Criteria:

* Documented history of any hypersensitivity of allergic reaction to any β-lactam antimicrobial.
* Confirmed or suspected infection with a pathogen known to be resistant to ceftriaxone.
* Confirmed or suspected respiratory tract infection attributed to sources other than CABP pathogens.
* Non-infectious causes of pulmonary infiltrates.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ceftaroline versus ceftriaxone in pediatric subjects age 2 months to <18 years with CABP requiring hospitalization | Between 1 and 50 days.
  Evaluate the safety and tolerability of IV administered ceftaroline fosamil in children with CABP. Summaries of AEs, SAEs, deaths, laboratory evaluations (hematology studies, comprehensive and metabolic panel), vital signs.

SECONDARY OUTCOMES:
Evaluate the efficacy of ceftaroline versus ceftriaxone in pediatric subjects ages 2 months to under 18 years with CABP. | Between 4 and 50 days
  * Clinical response by subject and by baseline pathogen at Study Day 4 in the Modified Intent-to-Treat (MITT) and Microbiological modified Intent-to Treat (mMITT) Populations
  * Clinical stability by subject and by baseline pathogen at Study Day 4 in the MITT and mMITT Populations
  * Clinical outcome at EOIV, EOT, and TOC in the MITT and Clinically Evaluable (CE) Populations
  * Clinical and microbiological outcomes by subject and by pathogen at TOC in the mMITT and Microbiologically Evaluable (ME) Populations
  * Clinical relapse at LFU in the MITT Population
  * Emergent infections in the mMITT Population
To evaluate the pharmacokinetics of ceftaroline in pediatric subjects ages 2 months to under 18 years. | Between 4 and 50 days
  Analyze concentrations of ceftaroline, ceftaroline fosamil (prodrug), and ceftaroline M-1 (inactive metabolite) in plasma, and, if available, in cerebrospinal fluid (CSF; if collected as part of standard of care).

CONTACTS AND LOCATIONS:
Locations (44):
- United States (13):
  - Investigational Site, Long Beach, California
  - Investigational Site, Oakland, California
  - Investigational Site, Orange, California
  - Investigational Site, San Diego, California
  - Investigational Site, Boston, Massachusetts
  - Investigational Site, Syracuse, New York
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Pittsuburg, Pennsylvania
  - Investigational Site, Memphis, Tennessee
  - Investigational Site, Houston, Texas
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, Morgantown, West Virginia
- Argentina (2):
  - Investigational Site, Capital Federal, Buenos Aires
  - Investigational Site, Córdoba, Córdoba Province
- Bulgaria (4):
  - Investigational Site, Plovdiv
  - Investigational Site, Rousse
  - Investigational Site2, Sofia
  - Investigational Site, Sofia
- Georgia (3):
  - Investigational Site2, Tbilisi
  - Investigational Site3, Tbilisi
  - Investigational Site, Tbilisi
- Greece (4):
  - Investigational Site, Athens, Attica
  - Investigational Site, Heraklion, Crete
  - Investigational Site, Thessaloniki, Macedonia
  - Investigational Site, Larissa, Thessaly
- Hungary (8):
  - Investigational Site, Gyula, Bekes County
  - Investigational Site, Ajka
  - Investigational Site, Budapest
  - Investigational Site, Nagykanisza
  - Investigational Site, Nyíregyháza
  - Investigational Site, Szeged
  - Investigational Site, Veszprém
  - Investigational Site, Zalaegerszeg
- Poland (3):
  - Investigational Site, Lublin
  - Investigational Site, Rzeszów
  - Investigational Site, Warsaw
- Spain (2):
  - Investigational Site, Madrid, Madrid
  - Investigational Site, Córdoba
- Ukraine (5):
  - Investigational Site, Donetsk
  - Investigational Site, Ivano-Frankivsk
  - Investigational Site, Kryvyi Rih
  - Investigational Site, Kyiv
  - Investigational Site, Zaporizhia

REFERENCES:
- [Derived] Cannavino CR, Nemeth A, Korczowski B, Bradley JS, O'Neal T, Jandourek A, Friedland HD, Kaplan SL. A Randomized, Prospective Study of Pediatric Patients With Community-acquired Pneumonia Treated With Ceftaroline Versus Ceftriaxone. Pediatr Infect Dis J. 2016 Jul;35(7):752-9. doi: 10.1097/INF.0000000000001159. PMID 27093162
- See also: sponsor website — http://www.cerexa.com